CLINICAL TRIAL: NCT02316496
Title: A Phase II Study of Cetuximab Rechallenge in Combination With Irinotecan in Advanced Metastatic Colorectal Cancer Without KRAS or NRAS or BRAF Mutation (All Wild Type) for Patients Pretreated With FOLFIRI and Cetuximab in First Line With Stopping Cetuximab for Progressive Disease After a Previous Response (Partial Response or Complete Response) and After Treatment With a Fluoropyrimidine, Oxaliplatin Plus Bevacizumab Regimen
Brief Title: Rechallenge of Cetuximab Combined With Irinotecan as Third-line Chemotherapy in Patients With Metastatic Colorectal Cancer - Phase II Study
Acronym: REGAIN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGAIN C13-2
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-01

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Cancer; Colorectal; Metastatic; Thrid-line; Irinotecan; Cetuximab
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label , single arm (Experimental): cetuximab - irinotecan until progression or unacceptable toxicity
  Interventions: Drug: cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: cetuximab — cetuximab 500mg/m²/ IV infusion, (q2w)
Drug: Irinotecan — Irinotecan 180mg/m², in 500ml NaCl 0.9% solution, 90 min IV infusion (q2w)

SUMMARY:
The main objective of this study is to evaluate the objective response rate at two months (complete disappearance of the disease and partial disappearance of the disease) obtained after administration of combination therapy with cetuximab and irinotecan in the patients with metastatic colorectal cancer.

Secondaries objectives will be assessed progression-free survival, overall survival, toxicity, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Histologically confirmed metastatic adenocarcinoma of the colon or rectum
* All Wild Type KRAS (exon 2 [codons 12-13], exon 3 [codons - 61]; exon 4 [codon 146]), NRAS (exon 2 [ codons 12-13] and exon 3 [codon 61) and BRAF (V600E) tumor ( local assessment performed either on primary tumor or metastasis)
* First line chemotherapy regimen with a fluoropyrimidine and Irinotecan (FOLFIRI) + cetuximab with initial partial or complete response and progressive disease (PD) with PD ≤ 6 weeks after the last administration of cetuximab
* Other line(s) of therapy(ies) including the following drugs: second line oxaliplatin based chemotherapy with fluoropyrimidines (5FU or capecitabine) + bevacizumab and eventually regorafenib (possible but not mandatory) and progression or limiting toxicity to the last therapy with a minimum of 4 months between last injection of cetuximab and inclusion in this study
* At least one measurable lesion ≥ 10 mm as assessed by CT-scan or MRI (Magnetic Resonance Imaging) according to RECIST v1.1 (All sites must be evaluated ≤ 28 days prior to the enrolment)
* Age ≥18 years
* World Health Organization (WHO) Performance status (PS) 0-2
* The patient has adequate organ function, defined as :

Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, hemoglobin ≥ 9 g/dL, and platelets ≥ 100 x 109/L.Total bilirubin ≤ 1.5 times upper limit of normal value (ULN), serum alkaline phosphatase level < 5 times ULN, Serum creatinine level <150μM/l

* For female patients of childbearing potential, negative pregnancy test within 7 days before starting the study drug
* Men and women are required to use adequate birth control during the study (when applicable) and until 6 months after the end of study treatment
* Registration in a national health care system (CMU included)

Exclusion Criteria:

* Previous chemotherapy other than adjuvant therapy with different combinations than those scheduled in first and second line treatment
* Presence of any KRAS, BRAF or NRAS mutation by allelic discrimination on tumor DNA
* Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiation of study treatment or a history of ventricular arrhythmia (treated or not)
* History or evidence of central nervous system metastasis (systematic CT-scan or MRI not mandatory if no clinical symptoms)
* Known allergy or hypersensitivity to cetuximab
* Previous or concurrent malignancy except for basal or squamous cell skin cancer, in situ carcinoma of the cervix, low-risk prostate cancer according to d'Amico classification or other solid tumors treated curatively and without evidence of recurrence for at least 5 years prior to the study
* Active or uncontrolled clinically serious infection
* Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness
* Other serious and uncontrolled non-malignant disease
* Pregnancy
* Breast feeding
* Treatment with any other investigational medicinal product within 28 days prior to study entry
* Known Gilbert's syndrome
* Concomitant administration of live, attenuated virus vaccine such as yellow fever vaccine
* Concomitant use with St John's Wort
* Chronic inflammatory bowel disease and/or Bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At 2 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 27 months
  Best response observed during investigational treatment combination. From the start of treatment until treatment failure
Disease control rate (DCR) | up to 27 months
  The proportion of patients with tumor response (Complete response or partial response) or tumor stabilization as best response during study treamtent
Progression-free survival (PFS) | up to 27 months
  Time from the date of inclusion to the date of the first progressive disease (RECIST criteria) or death (any cause)
Duration of response (DOR) | up to 27 months
  Only for patients with tumor response (complete reposne or partial response) , from first confirmed response to first observed progression (PD) or death due to PD during study treatment
Time to response (TTR) | up to 27 months
  Time from the date of inclusion to the date of the first confirmed CR or PR during study treatment
Time to progression (TTP) | up to 27 months
  Time from the date of inclusion to the date of the first obseved progression (PD), or death due to progression during the study treatment
Time to treatment failure (TTF) | up to 27 months
  Time from the date of inclusion to the date the decision was made to end the study treatment for any reason
Duration of stable disease (DoSD) | up to 27 months
  Only for patient with a stable disease (SD) as best response during the study treatment, from date of inclusion to the first observed progression (PD) or death due to progression
Overall survival (OS) | up to 27 months
  From the date of inclusion to the date of patient death, due to any cause, or to the last date the patient was known to be alive
Adverse Events (CTCAE v.4.03) | Up to 27 months
Quality of life | Up to 27 months
  Using EORTC Quality of Life Questionnaire - C30 (QLQ-C30) and the Dermatology Life Quality Index (DLQI ) questionnaires
Respose rate | up to 27 months
  RAS and BRAF status in circulating tumoral DNA
PFS | up to 27 months
  RAS and BRAF status in circulating tumoral DNA

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc GORNET, MD, Principal Investigator — Hôpital Saint Louis
Locations (20):
- France (20):
  - Hôpital Beaujon, Clichy
  - Centre hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Georges François Leclerc, Dijon
  - CHD Vendée, La Roche/ Yon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Européeen, Marseille
  - Institut Paoli-Calmettes, Marseille
  - CHU Caremeau, Nîmes
  - CHU Cochin, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Tenon, Paris
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Groupe hospitalier Public du Sud de l'Oise -site de Senlis, Senlis
  - Centre de radiothérapie - Clinique Sainte Anne, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpitaux du Léman, Thonon-les-Bains
  - CHU Tours - Hôpital Trousseau, Tours
  - Clinique Générale, Valence